CLINICAL TRIAL: NCT06422806
Title: A Randomized Phase III Trial of Doxorubicin + Pembrolizumab Versus Doxorubicin Alone for the Treatment of Dedifferentiated Liposarcoma (DDLPS), Undifferentiated Pleomorphic Sarcoma (UPS) and Related Poorly Differentiated Sarcomas
Brief Title: Measuring if Immunotherapy Plus Chemotherapy is Better Than Chemotherapy Alone for Patients With Aggressive Poorly Differentiated Sarcomas
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-06412; NCI-2023-06412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA7222 (Other: ECOG-ACRIN Cancer Research Group); EA7222 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-18; First posted 2024-05-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Dedifferentiated Liposarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IV Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Unresectable Dedifferentiated Liposarcoma; Unresectable Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Liposarcoma; Histiocytoma, Malignant Fibrous | interventions — Specimen Handling; X-Rays; Doxorubicin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (doxorubicin and pembrolizumab (Experimental): Patients receive doxorubicin IV over 3-10 minutes or up to 3 hours on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA scan, standard imaging scans and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab
- Arm B (doxorubicin) (Active Comparator): Patients receive doxorubicin IV over 3-10 minutes or up to 3 hours on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. At time of disease progression, patients may begin receiving pembrolizumab alone IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of additional progression or unacceptable toxicity. Patients also undergo ECHO or MUGA scan, standard imaging scans and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Diagnostic Imaging Testing — Undergo standard imaging scans
  Other Names: Diagnostic Imaging; Medical Imaging
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm A (doxorubicin and pembrolizumab

SUMMARY:
This phase III trial compares the effect of immunotherapy (pembrolizumab) plus chemotherapy (doxorubicin) to chemotherapy (doxorubicin) alone in treating patients with dedifferentiated liposarcoma (DDLPS), undifferentiated pleomorphic sarcoma (UPS) or a related poorly differentiated sarcoma that has spread from where it first started (primary site) to other places in the body (metastatic) or that cannot be removed by surgery (unresectable). Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's deoxyribonucleic acid (DNA) and may kill tumor cells. It also blocks a certain enzyme needed for cell division and DNA repair. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Adding immunotherapy (pembrolizumab) to the standard chemotherapy (doxorubicin) may help patients with metastatic or unresectable DDLPS, UPS or a related poorly differentiated sarcoma live longer without having disease progression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether the combination of doxorubicin and pembrolizumab will improve progression free survival (PFS) in UPS and related poorly differentiated sarcomas relative to doxorubicin alone.

II. To assess whether the combination of doxorubicin and pembrolizumab will improve PFS in DDLPS relative to doxorubicin alone.

KEY SECONDARY OBJECTIVE:

I. To assess whether the combination of doxorubicin and pembrolizumab versus (vs) the re-introduction of pembrolizumab in the doxorubicin alone arm at disease progression (i.e., upfront pembrolizumab vs second line pembrolizumab) improves overall survival (OS) in DDLPS and the UPS family of diseases.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability in each treatment arm. II. To quantify overall response rate (ORR) and durability of response (DOR) in each treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate the agreement between the central review and local Response Evaluation Criteria in Solid Tumors (RECIST) assessments for patients identified for central imaging review.

II. To compare PFS, OS, ORR and DOR of doxorubicin with or without pembrolizumab for all patients, combining the UPS and DDLPS patients together.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive doxorubicin intravenously (IV) over 3-10 minutes or up to 3 hours on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive doxorubicin IV over 3-10 minutes or up to 3 hours on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. At time of disease progression, patients may begin receiving pembrolizumab alone IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of additional progression or unacceptable toxicity.

Patients in both arms also undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan, standard imaging scans and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months in years 2-10.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have a confirmed histopathologic diagnosis of dedifferentiated liposarcoma (DDLPS), undifferentiated pleomorphic sarcoma (UPS) or a related poorly differentiated sarcoma. Because UPS can sometimes exist in a spectrum among related diagnoses, the following additional diagnostic will be allowed, but not limited to:

  * Pleomorphic sarcoma with inflammation or with limited areas of differentiation
  * Pleomorphic sarcoma with giant cells
  * Malignant fibrous histiocytoma (including storiform-pleomorphic and inflammatory subtypes)
  * Myxofibrosarcoma
  * Poorly differentiated sarcoma not otherwise specified (NOS)
  * Undifferentiated spindle cell sarcoma
  * Poorly differentiated spindle cell sarcoma NOS Any of these subtypes may have areas of focal myogenic differentiation
* Patient must have metastatic or unresectable sarcoma
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria:

  * Has achieved menarche at some point
  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. Contraception measures must continue for 6 months after the last dose of doxorubicin for patients of child bearing potential and for 3 months after the last dose of doxorubicin for male patients with partners of child bearing potential. Males with pregnant partners should use condoms during doxorubicin treatment and for at least 10 days after the last dose of doxorubicin. Contraception measures must also continue for 4 months after the last dose of pembrolizumab for patients of child bearing potential
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must have a left ventricular ejection fraction (LVEF) > 50% by either MUGA scan or echocardiogram obtained within 28 days prior to randomization
* Absolute neutrophil count (ANC) ≥ 1,500 cells/uL (must be obtained ≤ 7 days prior to protocol randomization)
* Platelets ≥ 75,000 cells/uL (must be obtained ≤ 7 days prior to protocol randomization)
* Total bilirubin < 1.2 mg/dL (must be obtained ≤ 7 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 × institutional upper limit of normal (ULN) (must be obtained ≤ 7 days prior to protocol randomization)
* Creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (must be obtained ≤ 7 days prior to protocol randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must not have a history of or active interstitial lung disease
* Patient must have measurable disease. Baseline imaging must include a chest computed tomography (CT). Imaging should be inclusive of all measurable and non-measurable disease and must be obtained within 28 days prior to randomization. Imaging must be available for uploading to Transfer of Images and Data (TRIAD)

  * NOTE: CT with (w/) contrast preferred, chest CT without contrast is acceptable, CT portion of positron emission tomography (PET) may be acceptable. Magnetic resonance imaging (MRI) is acceptable for measuring other sites of disease
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must not have had prior treatment with an anthracycline
* Patient must not have a diagnosis of clinically significant immunodeficiency or an autoimmune disorder requiring the patient to use systemic steroid chronically, or systemic steroids within 7 days prior to randomization
* Patient must not have a known history of active TB (Bacillus Tuberculosis)
* Patient must not have a known hypersensitivity to doxorubicin or pembrolizumab or any of their excipients
* Patients who have received prior chemotherapy, targeted small molecule therapy or radiation therapy must have recovered from the prior therapy at the time of randomization
* Patient must have recovered adequately from any prior major surgery prior to randomization
* Patient must not have had prior pericardial or mediastinal radiation
* Patient must not have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA4 agent
* Patient must not have an autoimmune or other disease that requires the use of daily corticosteroids of > 10 mg of prednisone (or equivalent). Patients who are on an active steroid taper at the time of randomization must finish prior to beginning study treatment. Patients who require inhaled or topical steroids are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to documented progression (per Response Evaluation Criteria in Solid Tumors version 1.1) or death from any cause without prior progression, up to 5 years
  Will be compared between the treatment arms (doxorubicin + pembrolizumab versus [vs] doxorubicin alone). The comparison of PFS between treatment arms will be done using a stratified (on Eastern Cooperative Oncology group performance status [0 vs 1]) log-rank test with a 2.5% type I error (1-sided). Will be analyzed separately for the undifferentiated pleomorphic sarcoma and related malignancies and for the dedifferentiated liposarcoma.

SECONDARY OUTCOMES:
Overall survival | From randomization to death, up to 5 years
  Will be compared between doxorubicin + pembrolizumab vs doxorubicin alone to test the strategy of upfront pembrolizumab vs second line pembrolizumab.

OTHER OUTCOMES:
Progression status | From randomization to documented progression (per RECIST version 1.1) or death from any cause without prior progression, up to 5 years
  Evaluated using Cohen's kappa coefficient.
Progression time | From randomization to documented progression (per RECIST version 1.1) or death from any cause without prior progression, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seth M Pollack, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (244):
- United States (235):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (6):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
- Puerto Rico (3):
  - Pan American Center for Oncology Trials LLC - Dorado, Dorado
  - Pan American Center for Oncology Trials LLC, San Juan
  - Pan American Center for Oncology Trials LLC - Ciudadela, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm